CLINICAL TRIAL: NCT02798081
Title: Virtual Reality Games for Elderly Socialization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Medicina do ABC (Other)
Responsible Party: Principal Investigator, Thaiany Pedrozo Campos Antunes, Master, Faculdade de Medicina do ABC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 52305215.3.0000.0082
Record Dates: First submitted 2016-05-31; First posted 2016-06-14 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Aged
Keywords: augmentative and alternative communication; social inclusion; serious games; Information and communication technologies
MeSH Terms: conditions — Social Inclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm study (Experimental): A minimum of 46 elderly, students of a informatics course, will participate in the study. Initially, the students will have 8 usual informatics classes in the institution where they were enrolled spontaneously. Then, during the next 8 classes (from class 9 to class 16) they will practice 10 minutes of virtual reality games, as part of the class.
  Interventions: Behavioral: Single arm study

INTERVENTIONS:
Behavioral: Single arm study — In Step 1 the elderly will participate of eight conventional computer classes which they were spontaneously enrolled. In Step 2, 10 minutes of the next eight classes will be used to practice serious games using virtual reality, using physical interface (keyboard or mouse).
  Other Names: practicing virtual reality games

SUMMARY:
A minimum of 23 people aged 60 years and older, of both sexes, from an informatics course for beginners will participate in the study. The evaluation will consist mainly in answering two validated questionnaires on socialization, the short Social and Emotional Loneliness Scale for Adults (SELSA-S) and short-form UCLA Loneliness Scale (ULS-6). Reaction time and performance will also be measured by three virtual reality games, namely Reaction Time, Random and Moviletrando. All this evaluation will be repeated in three moments: T0 - at baseline; T1 - after 8 conventional informatics classes and; T2 - after 8 informatics classes which includes 15 minutes for practicing virtual reality games.

DETAILED DESCRIPTION:
Background: The use of new Technologies, such as the resources of augmentative and alternative communication (AAC), appears as a valuable tool to promote socialization in many groups of people. Serious games with virtual reality are an example of these resources and might bring benefits also to the elderly population, allowing an enjoyable and safe interaction that uses various sensorial stimuli. The purpose of this study protocol is to evaluate the effects of practicing virtual reality games on elderly socialization.

Method/Design: It will be an experimental, prospective longitudinal study which will use serious games with virtual reality to improve the socialization of elderly people. A minimum of 23 people aged 60 years and older, of both sexes, from an informatics course for beginners will participate in the study. The evaluation will consist mainly in answering two validated questionnaires on socialization, the short Social and Emotional Loneliness Scale for Adults (SELSA-S) and short-form UCLA Loneliness Scale (ULS-6). Reaction time and performance will also be measured by three virtual reality games, namely Reaction Time, Random and Moviletrando. All this evaluation will be repeated in three moments: T0 - at baseline; T1 - after 8 conventional informatics classes and; T2 - after 8 informatics classes which includes 15 minutes for practicing virtual reality games.

Discussion: This study will determine whether the practice of virtual reality games in addition to the usual informatics classes contributes to elderly socialization. The evolution in socialization, the evolution of reaction time and performance in virtual reality games and the correlation of motor learning to socialization will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* people aged over 60 years;
* both sexes
* spontaneously enrolled in the informatics beginner class for seniors of the Center of Reference for Elderly (CRI) in Ribeirão Pires

Exclusion Criteria:

* Less than 75% of frequency in the classes between the assessments;
* do not completion of the three moments of assessment;
* having motor impairment of the upper limbs or cognition impairment,which prevents them to practice the games.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Socialization assessed by SELSA-S | up to 10 weeks
  Improvement on self-perceived loneliness, representing the socialization level of the elderly, comparing baseline to the first 8 usual computer classes and after the 8 classes with virtual reality games. This will be verified through a decrease in the score of SELSA-S.
  SELSA-S has 15 items, scoring up to 7 in each, 105 in total.

SECONDARY OUTCOMES:
time of response during the practise of virtual reality games as assessed by TRT, Random and Moviletrando | up to 10 weeks
  It's expected to have a decrease in time of response during the practise of virtual reality games. It will be recorded by the softwares of the games: Time response (TRT), Random and Moviletrando

CONTACTS AND LOCATIONS:
Overall Officials: Thaiany Antunes, Master, Principal Investigator — Faculdade de Medicina do ABC
Locations (1):
- Faculdade de Medicina do ABC, Santo André, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Antunes TPC, Oliveira ASB, Crocetta TB, Antao JYFL, Barbosa RTA, Guarnieri R, Massetti T, Monteiro CBM, Abreu LC. Computer classes and games in virtual reality environment to reduce loneliness among students of an elderly reference center: Study protocol for a randomised cross-over design. Medicine (Baltimore). 2017 Mar;96(10):e5954. doi: 10.1097/MD.0000000000005954. PMID 28272198